CLINICAL TRIAL: NCT04018079
Title: Left Ventricular Dysfunction Post Surgical Patent Ductus Arteriosus Ligation in Children: Predictor Factors Analysis
Brief Title: Left Ventricular Dysfunction Post-surgical Patent Ductus Arteriosus Ligation in Children: Predictor Factors Analysis
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Bary Ahmed Ibrahim, Associate professor, South Valley University
Other Study IDs: South Valley University 1513
Record Dates: First submitted 2019-06-03; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Congenital Heart Disease in Children
Keywords: PDA; Echo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

PDA is viewed as a standout amongst the most widely recognized congenital heart defects in children and its closure is responsible for many hemodynamic changes that require intervention and care.

Methods:

A retrospective study included fifty children with isolated PDA treated by surgical ligation from June 2015 to June 2018. Their mean age was 15.78 ± 7.58 months and 72% were females. The LV dimensions and systolic function were assessed by two-dimensional echocardiography pre PDA ligation. The mean duct size was 4.08 ± 1.25 mm.

DETAILED DESCRIPTION:
Methods:

Study population Fifty children with PDA, for whom surgical PDA ligation was done from June 2015 to June 2018. All cases were operated in cardiothoracic surgery department and were followed up by cardiothoracic surgeons and paediatricians at cardiac surgery ICU, Qena University Hospital. Their mean age at intervention was 15.78 ± 7.58 months, body surface area (BSA) 0.43±0.03 and 32 (72%) were females. The mean duct diameter was 4.08 ± 1.25 mm. The study conforms to the ethical standards of the Helsinki Declaration and approval was obtained from the institutional ethics committee of Qena Faculty of Medicine.

Surgical technique PDA ligation was performed under general anaesthesia after pre-operative anaesthetic evaluation. After single endotracheal tube anaesthesia induction; children were placed on the right lateral recumbent position fixed with adhesive plaster and a pad under the chest, the left arm raised above the head. A left mini-thoracotomy incision is done parallel to the medial border of the scapula and entrance to the thoracic cavity was via the third or fourth intercostal space. Cautiously, the ductus is identified and dissected carefully. Then it was doubly ligated with silk ligature (2/0 or 0). An intercostal tube inserted during operation and removed within 48 hours if no drainage presents.

Descriptive statistical analysis Data were arranged and analyzed utilizing Version 20 of the SPSS program (Statistical Package for Social Sciences). Continuous variables were compared using the Student paired t-test and are expressed as mean values ± standard deviation. Pearson Chi-Square tests were used to detect differences among groups for categorical variables. The relationship between PDA size and changes in echocardiographic parameters was verified using the Pearson linear correlation and the linear regression analysis. P-value of <0.05 was considered of significance.

ELIGIBILITY:
Inclusion Criteria:

* All cases had clinical as well as echocardiographic proof of hemodynamically critical PDA.

Exclusion Criteria:

* Patients with silent PDA.
* irreversible pulmonary vascular disease.
* those who had associated hemodynamically significant congenital heart disease (CHD).

Ages: 8 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All cases were operated in cardiothoracic surgery department and were followed up by cardiothoracic surgeons and paediatricians at cardiac surgery ICU, Qena University Hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Comparison between the echocardiographic changes before PDA ligation to the follow up changes at one day, one month and six months post PDA ligation. | echocardiography was done before PDA ligation; and follow up at one day, one month and six months post ligation.
  the echocardiographic data included: The LV end-diastolic dimension (LVEDd) in mm, LV end-systolic dimension (LVESd) in mm, PDA size in mm, left atrial to aortic diameter ratio (LA/Ao ratio), EF % and FS %

SECONDARY OUTCOMES:
identification of the preoperative predictor factors of LV dysfunction following PDA surgical ligation in children | all data were collected pre ligation; at one day, one month and six months post ligation
  we classified our patients into two gatherings as indicated by FS % based on a definition of LV systolic dysfunction; group I with FS ≤ 29% and group II with FS > 29%.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdel-Bary M, Abdel-Baseer KA, Abdel-Latif AF, Abdel-Naser MA, Nafie M, Eisa KM. Left ventricular dysfunction postsurgical patent ductus arteriosus ligation in children: predictor factors analysis. J Cardiothorac Surg. 2019 Sep 18;14(1):168. doi: 10.1186/s13019-019-0990-z. PMID 31533759